CLINICAL TRIAL: NCT04222738
Title: Short Term Cardiovascular Effects of Zingiber Officinale as add-on Therapy in a Population of Type 2 Diabetes Individuals
Brief Title: The Cardiovascular Effects of Ginger (Zingiber Officinale) in Patients With Type II Diabetes Mellitus
Acronym: GINOFF1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: NGATI Denetria NYONGA, Dr (Unknown); SOBNGWI Eugène, Pr (Unknown); MBANYA Jean Claude, Pr (Unknown)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ginger and type 2 diabetes
Record Dates: First submitted 2019-03-05; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Benefits of Zingiber Officinale Roscoe in Patients With Type 2 Diabetes Mellitus Before and After 6 Weeks of add-on Therapy
Keywords: Diabetes mellitus; Diastolic function; Blood pressure; Zingiber officinale
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-randomized single-arm of GINOFF1 (Experimental): Non-randomized single-arm clinical trial with a before and after design. The study population consisted on all type 2 diabetes mellitus (T2DM) patients with a target population of T2DM patients with HbA1c between 42 to 64mmol/mol (6-8%) with no change in anti-diabetic treatment during the last three months, previous the study.
  The intervention consisted on the administration of Zingiber officinale Roscoe extracts, at a daily dose of 2g/day (equivalent overall daily dose of extract in simple powdered form) for a period of 6weeks. The extracts were given as capsules, either one capsule three times per day (1 capsule x 3 / day) and after meals. Each capsule contains 399mg of pure Zingiber officinale Roscoe extracts.
  Interventions: Dietary Supplement: GINOFF1

INTERVENTIONS:
Dietary Supplement: GINOFF1 — The intervention lasted for six weeks and consisted of the administration of powdered ginger extracts in the form of capsules at a dose of 2g/day.

SUMMARY:
The aim of the study was the evaluation of cardiovascular benefits of Zingiber officinale Roscoe in patients with type 2 diabetes mellitus before and after 6 weeks of add-on therapy.

DETAILED DESCRIPTION:
the investigators performed a non-randomized single-arm clinical trial with a before and after design, carried out from December 2016 and May 2017.

Intervention consisted of the administration of powdered ginger extracts in the form of capsules at a dose of 2g/day, for a period of 6 weeks. Before and after intervention, the following were done by the participants: bioelectrical impedance analysis (BIA), blood pressure measurements, fasting blood sugar, HbA1c, lipid profiles, liver function tests, kidney function tests and full blood counts. These were followed by morphological workup including Electrocardiograms (ECGs), transthoracic heart ultrasounds and Ambulatory Blood Pressure Measurements (ABPM), also done before and after intervention.

Clinical evaluation with fasting blood sugar control and blood pressure controls were done at day 21 for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Known T2DM patients aged above 21years
* No change in anti-diabetic medication during the last three months.
* HbA1c between 42 to 64mmol/mol (6-8%).

Exclusion Criteria:

* Patient already on ginger supplementation or other herbal medication
* Drugs that could interact with ginger or whose effects may be amplified such as NSAIDS, corticosteroids and anticoagulants like heparin or warfarin, as far back as 1 month before study.
* Cardiac, renal disease and liver pathologies
* Heartburn or peptic ulcer disease
* Sensitivity, intolerance or allergy to ginger
* Discontinued intervention
* Withdrawal of consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Variation of mitral E' velocity | 6 weeks
  The mitral E' velocity is one of the methods for evaluating diastolic function.

SECONDARY OUTCOMES:
Variation of transmitral flow parameters such as E velocity | 6 weeks
  E (early diastolic filling velocity)
Variation of blood pressure. | 6 weeks
  Change in systolic and diastolic blood pressure by using ABPM (mmHg)
Variation of weight loss | 6 weeks
  Change in weight (Kgs)
Variation of HbA1c | 6 weeks
  Change in HbA1c (%)
Variation of lipid profile. | 6 weeks
  Change of triglycerides, LDL cholesterol, HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nadege NGANOU-GNINDJIO, MD, MAS, Principal Investigator — Yaounde Central Hospital; Eugene SOBNGWI, Professor, Study Director — Yaounde Central Hospital; Jean Claude MBANYA, Professor, Study Chair — Yaounde Central Hospital
Locations (1):
- Yaounde Central Hospital, NAtional Obesity Center, Yaoundé, Cameroon

REFERENCES:
- [Derived] Nganou-Gnindjio CN, Ngati Nyonga D, Wafeu GS, Nga EN, Sobngwi E. Cardiometabolic effects of ZingiberOfficinale Roscoe extracts in Type 2 diabetic Cameroonians patients after six weeks of add-on Therapy : A single clinical-arm trial. Ann Cardiol Angeiol (Paris). 2022 Jun;71(3):160-165. doi: 10.1016/j.ancard.2021.09.010. Epub 2022 Jan 14. French. PMID 35039142